CLINICAL TRIAL: NCT03594032
Title: Prevalence and Clinical Characteristics of Patients With Bronchiectasis With Comorbid Nontuberculous Mycobacteria Among Middle-aged and Old Women
Brief Title: Prevalence and Characteristics of Patients With Bronchiectasis Comorbid Nontuberculous Mycobacteria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bin Cao (Other)
Responsible Party: Sponsor-Investigator, Bin Cao, Clinical professor, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: 2018-62-K46
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Bronchiectasis; Non-tuberculous Mycobacterial
Keywords: bronchiectasis; NTM infections; Middle-aged and old women
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to Understand the prevalence of non-tuberculous mycobacterial(NTM) infections in the middle-aged and old women patients with bronchiectasis in Mainland China, and explore the characteristics of patients with bronchiectasis comorbid NTM.

DETAILED DESCRIPTION:
The development of bronchiectasis is closely related to chronic infection of pathogenic microorganisms .Bronchiectasis and nontuberculous mycobacterial (NTM) infections are inextricably linked Pathophysiologically. But the incidence rate and characteristics of NTM infections among patients with bronchiectasis remains unclear in mainland China.

In this study, we will collect data of participants about demographic ,co-morbidities ,spirometry, mMRC score ,exacerbation history, QOL-B questionnaire, aetiology, spirometry , HRCT(or CT) scan ,results of microbiology samples and treatments, collect three consecutive sputum(or induced sputum) samples to smear, bacteria culture, acid-fast stain, mycobacterium cultivation and identification, drug susceptibility testing of nontuberculous mycobacteria.To estimate the prevalance of non-tuberculous mycobacterial(NTM) infections in Middle-aged and old women patients with bronchiectasis in northern China. To analyze clinical manifestations and microbiological characteristics of patients with bronchiectasis comorbid NTM infections By 16SRNA and gene sequencing.

In addition, A cross-sectional investigation about lung function and clinical data will be done among patients who have confirmed bronchiectasis with NTM from February 2017 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Middle-aged and old women who are > or = 50 years of age
2. Patients meet the criteria of bronchiectasis

Exclusion Criteria:

1. Cystic fibrosis
2. After organ transplantation
3. Activity tumor (malignant solid tumor and blood system tumor)
4. Pulmonary interstitial fibrosis with bronchus dilation
5. Allergic bronchopulmonary aspergillosis
6. Diffuse panbronchiolitis
7. Patients refused to sign the informed consent
8. Patients unable to return sputum specimens

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 216 patients with bronchiectasis who meet the below inclusion criteria will be re cruited in China-Japan Friendship Hospital in Beijing,China.
Sampling Method: Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
NTM infection rates | 24 months afer enrolled participants
  NTM infection rates in Middle-aged and old women patients with bronchiectasis in northern China

SECONDARY OUTCOMES:
clinical characteristics of patients with bronchiectasis comorbid NTM infections | 24 months afer enrolled participants
  clinical manifestations of patients with bronchiectasis comorbid NTM infections
microbiological characteristics of patients with bronchiectasis comorbid NTM infections | 24 months afer enrolled participants
  microbiological characteristics of patients with bronchiectasis comorbid NTM
Drug resistance of NTM | 24 months afer enrolled participants
  drug susceptibility testing outcomes of nontuberculous mycobacteria from sputum samples

CONTACTS AND LOCATIONS:
Overall Officials: Ben Cao, MD, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yin H, Gu X, Wang Y, Fan G, Lu B, Liu M, Wang C, Cao B, Wang C. Clinical characteristics of patients with bronchiectasis with nontuberculous mycobacterial disease in Mainland China: a single center cross-sectional study. BMC Infect Dis. 2021 Dec 6;21(1):1216. doi: 10.1186/s12879-021-06917-8. PMID 34872515